CLINICAL TRIAL: NCT07279090
Title: Spatiotemporal Single-cell Atlas of Peri-implant Soft Tissue Healing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stomatological Hospital Affiliated with Fujian Medical University (Other)
Responsible Party: Principal Investigator, Cheng Hui, Professor of Prosthodontics, Stomatological Hospital Affiliated with Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20250829
Record Dates: First submitted 2025-09-16; First posted 2025-12-12 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Peri-implant Soft Tissue Healing
Keywords: Peri-implant soft tissue healing; scRNA-seq

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healing Abutment Gingival Healing Post-Implantation (Experimental)
  Interventions: Procedure: Healing Abutment Gingival Healing Post-Implantation

INTERVENTIONS:
Procedure: Healing Abutment Gingival Healing Post-Implantation — The healing process of peri-implant soft tissues will be studied using a micro healing abutment (2 mm), which will be placed at least three months after implant Stage I surgery. Gingival tissue samples will then be collected at Day 4, Week 2, Week 4, and Week 8-10. At each time point, a circular incision around the micro abutment will be made using a circular punch, and the gingival tissue together with the abutment will be retrieved under local anesthesia. After sampling, the micro abutment will be replaced with a formal healing abutment to maintain healing. Samples will undergo single-cell RNA sequencing (scRNA-seq) to characterize cell types, gene expression changes, and regulatory pathways involved in soft tissue repair. Additional tissues will be used for spatial transcriptomics (ST) and histological staining.

SUMMARY:
This study aims to explore the dynamic changes in different cell types and their molecular regulatory mechanisms during the healing process of peri-implant soft tissues, using single-cell RNA sequencing (scRNA-seq) and spatial transcriptomics (ST).

The research will focus specifically on the healing of soft tissues around dental implants in human subjects with the use of a healing abutment. Participants in the healing abutment group will have a micro healing abutment placed immediately after implant placement.

Tissue samples will be collected at various time points (Day 4, Day 14, and Day 70) to construct a detailed single-cell map of the healing process.

Spatial transcriptomics will be integrated to preserve tissue architecture, enabling the identification of the spatial distribution of different cell types and their interactions within the peri-implant microenvironment.

This combined approach will allow for a comprehensive characterization of cellular interactions, spatial gene expression patterns, and regulatory networks specific to healing abutments.

The goal is to identify key regulatory factors that could improve peri-implant soft tissue healing and help prevent peri-implantitis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* Healthy individuals without chronic medical conditions or severe systemic diseases
* Able to comply with study requirements (e.g., follow-up visits)
* No history of periodontal disease or active infection
* Already completed four or more implant placements in the posterior tooth region
* Adequate gingival thickness to allow for sampling and proper healing

Exclusion Criteria:

* Individuals with systemic conditions that affect wound healing (e.g., diabetes, immunosuppressive therapy)
* Smoking or alcohol abuse
* Pregnant or breastfeeding women
* History of severe allergic reactions to implant materials
* Participation in another clinical study at the same time

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome 1: Differentially Expressed Genes (DEGs) in Peri-implant Soft Tissues | Day 4, Week 2, Week 4 and Week 8-10 post-implantation.
  Number of genes significantly differentially expressed between experimental groups, determined by single-cell RNA sequencing (scRNA-seq) analysis (FDR < 0.05).
  Unit of Measure: Number of genes.
Cell Type Composition in Peri-implant Soft Tissues | Day 4, Week 2, Week 4, and Week 8-10 post-implantation.
  Proportion (%) of each annotated cell type identified by scRNA-seq based on canonical marker expression.
  Unit of Measure: Percentage of total cells (%)
Enriched Biological Pathways | Day 4, Week 2, Week 4, and Week 8-10 post-implantation
  Number of significantly enriched Gene Ontology (GO) terms and KEGG pathways identified from DEGs (FDR < 0.05).
  Unit of Measure: Number of enriched terms/pathways
Ligand-Receptor Interaction Strength | Day 4, Week 2, Week 4, and Week 8-10 post-implantation
  Mean interaction score of ligand-receptor pairs identified among annotated cell types using CellPhoneDB (or equivalent computational tool).
  Unit of Measure: Interaction score (arbitrary units)
Spatial Gene Expression Patterns | Day 4, Week 2, Week 4 and Week 8-10 post-implantation.
  Localization and expression intensity of selected DEGs across tissue regions determined by the 10x Genomics Visium platform.

SECONDARY OUTCOMES:
Histological Tissue Morphology | Day 4, Week 2, Week 4 and Week 8-10 post-implantation.
  Assessment of epithelial continuity, connective tissue organization, and inflammatory cell infiltration in peri-implant soft tissues by hematoxylin and eosin (H&E) staining. Each parameter will be semi-quantitatively scored on a standardized histological scale (0-3), where 0 = none, 1 = mild, 2 = moderate, and 3 = severe.
Immune and Stromal Cell Quantification | Day 4, Week 2, Week 4 and Week 8-10 post-implantation.
  Quantification of immune cells (e.g., CD68⁺ macrophages, CD3⁺ T lymphocytes) and stromal cells (e.g., fibroblast-related markers) by immunohistochemistry (IHC). Mean positive cell count per high-power field (HPF) will be calculated from representative sections.
Junctional Epithelium Length | Day 4, Week 2, Week 4, and Week 8-10 post-implantation.
  Measurement of junctional epithelium length along the implant surface using histological sections and digital image analysis software.
  Unit of Measure: Length (µm)
Basement Membrane Protein Expression | Day 4, Week 2, Week 4, and Week 8-10 post-implantation.
  Immunohistochemical detection of Laminin-332 and related basement membrane proteins indicating epithelial attachment integrity. The percentage of positive staining area will be quantified using image analysis software.
  Unit of Measure: Percentage of positive area (%)

CONTACTS AND LOCATIONS:
Locations (1):
- School and Hospital of Stomatology, Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided
Taking into account factors such as the needs of subsequent research, the final decision has not yet been made.